CLINICAL TRIAL: NCT06296199
Title: Music, Virtual Reality and Mental Health of Inpatients in the Intensive Functional Rehabilitation Unit and Patients in the IUGM Geriatric Outpatient Clinic: Pilot Clinical Trial
Brief Title: Music, Virtual Reality for Patients in IUGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal (Other Government)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, director of AgeTeQ Lab at CRIUGM, Centre integre universitaire de sante et de services sociaux du Centre-Sud-de-l'Île-de-Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-2064
Record Dates: First submitted 2024-02-22; First posted 2024-03-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Aging; Disorder, Neurologic
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): participants will listen to and watch a concert of musicians playing classical music through a VR headset
  Interventions: Other: VR
- Control (Active Comparator): participants will simply listen to the concert through headphones
  Interventions: Other: Music only

INTERVENTIONS:
Other: VR — The participant will be seated comfortably in an armchair. The intervention will last 15 minutes. It will take place once.
  This group's intervention will be to watch and listen with VR headphones to a concert by a group of musicians playing music.
  Arms: Intervention
Other: Music only — The participant will be seated comfortably in an armchair. The intervention will last 15 minutes. It will take place once.
  This group's intervention will be to listen with conventional headphones to a concert by a group of musicians playing music.
  Arms: Control

SUMMARY:
Promoting good care, well-being and quality of life for geriatric patients is a long-standing initiative in Quebec, and one in which the Institut Universitaire de Gériatrie de Montréal (IUGM) has always been a leader. For example, the IUGM played a major role in drafting the reference framework for the AAPA (approach adapted to the needs of the elderly), which was introduced by the Ministère de la Santé et des Services Sociaux in 2011. The investigator propose to continue this work by focusing in this project on the development of a new intervention aimed at the well-being and quality of life of geriatric patients and based on music and VR.

Thee investigator hypothesize (1) that a VR headset-based intervention based on listening to and observing a concert of musicians playing classical music is feasible for patients hospitalized at the IUGM's URFI and in patients attending the geriatric outpatient clinic, and (2) that this intervention can improve their mental health - i.e. their positive emotions, well-being and quality of life - and reduce their anxiety.

ELIGIBILITY:
Inclusion Criteria:

* be hospitalized at the URFI of the IUGM, or being a patients attending the geriatric outpatient clinic
* be 60 years of age or older,
* not have an acute intercurrent pathology in the week preceding the procedure and during the two days of the procedure,
* have no psycho-behavioural disorders,
* no major neurocognitive disorder at a severe stage,
* no severe visual or hearing impairment,
* no vestibular balance disorders,
* give written consent to participate in the study.

Exclusion Criteria:

* Participate in another concurrent experimental clinical study, to avoid interference with our study.
* Do not understand written or spoken French or English. The participants are French and/or English speakers, and the questionnaires are only available in these 2 languages.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-10-23 (Actual); Study Completion 2024-10-23 (Actual)

PRIMARY OUTCOMES:
Feasability | 6 months
  To determine if investigator is able to recruit 80 patients in 6 months, with a consent rate of 80% or more and less than 20% of withdrawal

SECONDARY OUTCOMES:
Emotions variation | 1 day
  To quantify and compare variations in Visual Analog Mood Scales (VAMS) score between the intervention group (listening to and watching musicians with VR headphones) and the control group (listening to music with headphones).
  This scale examines 8 emotions represented by ideogrammatic icons. It contains 2 positive emotions (happy and energetic) and 6 negative emotions (scared, confused, sad, angry, tired, tense). Each emotion is linked to a neutral face by a line. Participants will be asked to place a mark on the line at the point that represents the intensity of the emotion they are feeling. The distance in millimetres from the neutral face corresponds to the score (e.g., the further away from the neutral face, the greater the emotion). A higher positive emotion score means the participant feels better, and a higher negative emotion score means the patient feels worse.
Affect variation | 1 day
  To quantify and compare variations in scores on Positive and negative Affect schedule (PANAS) between the intervention group (listening to and watching musicians with VR headphones) and the control group (listening to music with headphones).
  This positive and negative affectivity scale is a questionnaire designed to measure the valence and activation (i.e. intensity) of a person's affects. It comprises two scales. The first measures positive affect, the second negative affect. Each scale comprises 10 items, for a total of 20. Scores range from 10 to 50 for the negative affect score and from 10 to 50 for the positive affect score, respectively, with a low score representing the lowest levels of negative affect, and a high score representing high levels of positive affect. A high negative affect score reveals psychological distress involving a variety of unpleasant emotions, while a low score reflects calm and serenity.
Well-Being Variation | 1 day
  To quantify and compare variations in scores on Warwick Edinburgh mental well-being scale measuring well-being between the intervention group (listening to and watching musicians with VR headphones) and the control group (listening to music with headphones).
  This scale is made up of 14 positively worded items and produces scores ranging from 14 (i.e. no well-being) to 70 (i.e. complete well-being).
Quality of life variation | 1 day
  To quantify and compare variations in scores on Eq-5D scale measuring quality of life between the intervention group (listening to and watching musicians with VR headphones) and the control group (listening to music with headphones).
  This test is a standardized measure of health status developed by the EuroQol group to provide a simple, generic measure of health for clinical and economic evaluation. It provides a simple descriptive profile and a single index value for health status. The EQ-5D consists of two parts: (1) a five-question questionnaire with a score per question ranging from 1 (i.e. no problem) to 5 (i.e. a more serious problem), (2) and a visual analog scale indicating how good or bad the participant's health is. This scale is numbered from 0 (i.e. the worst health the participant can imagine) to 100 (i.e. the best health the participant can imagine).
Anxiety variation | 1 day
  To quantify and compare variations in scores on General Anxiety Disorder - 7 scale measuring anxiety between the intervention group (listening to and watching musicians with VR headphones) and the control group (listening to music with headphones).
  This is a 7-item scale (each item is rated on a Likert scale ranging from "not at all" to "almost every day"). The maximum score is 21, and the higher the score, the greater the anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- CRIUGM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No